CLINICAL TRIAL: NCT01425788
Title: Comparison of Different Up-dosing Schedules With Osiris Phleum Pratense
Acronym: Osiris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Ergomed (Industry); ACM Pivotal Global Central Laboratory (Industry); Brecon Pharmaceuticals Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OS-G-01
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Rhino-conjunctivitis
Keywords: Grass pollen induced allergic rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Osiris Phleum pratense - Group A (Active Comparator): Group A up-dosing schedule from 1IR (index of Reactivity) /day to 240 IR/day in 11 days and thereafter 300 IR/day in 19 days.
  Day 1-6: 1,2,4,6,8,10 IR/day Day 7-11: 30, 60, 120, 180, 240 IR/day Day 12-30: 300 IR/day
  Interventions: Biological: Osiris Phleum pratense
- Osiris Phleum pratense - Group B (Active Comparator): Group B Up-dosing schedule:
  Day 1-5: 50 IR/day Day 6-10: 150 IR/day Day 11-30: 300 IR/day
  Interventions: Biological: Osiris Phleum pratense
- Osiris Phleum pratense - Group C (Active Comparator): Group C up-dosing schedule:
  Day 1-10: 50 IR/day Day 11-20: 150 IR/day Day 21-30: 300 IR/day
  Interventions: Biological: Osiris Phleum pratense

INTERVENTIONS:
Biological: Osiris Phleum pratense
  Arms: Osiris Phleum pratense - Group A
Biological: Osiris Phleum pratense
  Arms: Osiris Phleum pratense - Group B
Biological: Osiris Phleum pratense
  Arms: Osiris Phleum pratense - Group C

SUMMARY:
The purpose of this trial is to investigate the tolerability of Osiris Phleum pratense used with 2 simplified up-dosing schedules compared to the up-dosing schedule used in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before entering the trial
* Male or female >/= 18 years at visit 1
* A clinically relevant history of grass pollen induced allergic rhinoconjunctivitis (moderate to severe) and having received symptomatic treatment during grass pollen season 2010 and 2011
* Positive skin prick test response (wheal diameter >/= 3mm) to Phleum pratense
* Positive specific IgE against Phleum pratense (>/= 0,70KUL / class 2)
* Female subjects of childbearing potential must have a negative pregnancy test and be willing to practice appropriate contraceptive methods until Visit 4
* Subjects willing and able to comply with trial protocol regimen

Exclusion Criteria:

* Subjects included in another protocol (treatment intervention and/or investigational medicine product) or having participated in another clinical trial within 30 days prior to visit 1
* A clinically relevant history of symptomatic seasonal allergic rhinoconjunctivitis caused by an allergen (e.g. hazel, alder, birch, ash) to which the subject will be exposed during the 30-day treatment period.
* A clinically relevant medical history of symptomatic perennial allergy to allergen(s) to which the subject is regularly exposed (e.g. cat, house dust mites).
* Known sensitization (history of positive SPT) to food allergens with oral allergy syndrome
* Uncontrolled asthma (in accordance with GINA guidelines) within the last 12 months
* FEV < 60% of predicted within the last 12 months
* Severe asthma exacerbation(s) within the last 12 months
* A clinically relevant chronic disease (>/= 3 months) (e.g fibrosis, malignancy, type 1 diabetes mellitus, malabsorption or malnutrition, renal or hepatic insufficiency)
* Malignancy or systemic disease affecting the immune system (e.g. autoimmune disease, immune complex disease or immune deficiency disease)
* Inflammatory conditions in the oral cavity with severe symptoms such as oral lichen planus with ulcerations or severe oral mycosis or dental extraction at randomisation
* Medical history of recurrent urticaria or atopic dermatitis during the last 2 years
* Currently receiving treatment preventing the initiation of SIT (e.g. tricyclic antidepressants, mono amine oxidase inhibitors (MAOIs) and catechol-O-methyl transferase inhibitors (COMT inhibitors))
* History of allergy, hypersensitivity, or intolerance to the excipients of the investigational medicinal product
* Being immediate family of the investigator or trial staff, defined as the investigator's / staff's spouse, parent, grandparent, child or grandchild
* History of drug induced (incl. immunotherapy) facial angioedema (including experience of Quincke oedema) or a family (parents or siblings) history of hereditary angioedema
* Anticipated use of any prohibited medication within the specified time windows as defined in the protocol
* Previous treatment by immunotherapy with grass pollen for more than one month within the last 5 years
* Any clinically significant condition or situation, other than the condition being studied, that in the opinion of the investigator would interfere with the trial evaluations or optimal participation
* History of anaphylaxis with cardio respiratory symptoms (e.g. food allergy, drugs or an idiopathic reaction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Tolerability based on reporting of adverse events | An average of 42 days per subject
  Recording of adverse events are performed during the entire trial period, from screening to final follow-up contact.

SECONDARY OUTCOMES:
Subject satisfaction | Measured at "End of treatment/end of trial Visit"
  To compare the subjects' satisfaction of the different dosing schedules at end of the trial (after 30 days of treatment with trial medication).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Prof.med, Principal Investigator — Uniwersytecki Szpital Kliniczny Nr1, Lodz, Poland
Locations (1):
- Poradnia Alergologii i Chorob Pluc Uniwersyteckiego Szpitala Klinicznego Nr1 im. N. Barlickiego w Lodzi, Lodz, Poland